CLINICAL TRIAL: NCT06516562
Title: Demographic, Clinical, Biological, Treatment Characteristics and Cardiovascular Events of Patients With Heart Failure in Vietnam: a Multicenter Prospective Observational Study
Acronym: MCR-HF
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Other Study IDs: 43/2024/HĐ-ĐHYD
Record Dates: First submitted 2024-07-17; First posted 2024-07-24 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Heart Failure With Mid Range Ejection Fraction
Keywords: Patient registry; Heart failure; Prospective Observational Study; Demographic; Treatment characteristics; Prognosis; MACE
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart failure with reduced or mildly reduced ejection fraction
  Interventions: Drug: Optimal treatment

INTERVENTIONS:
Drug: Optimal treatment — Optimal treatment using current National Guidelines for the diagnosis and treatment of chronic heart failure

SUMMARY:
Describe the clinical characteristics, paraclinical features, and treatment during hospitalization, as well as at 1, 3, and 12 months post-discharge, of heart failure patients at selected cardiovascular centers in Vietnam.

DETAILED DESCRIPTION:
Study Design: Prospective cohort study

Study Subjects: Patients discharged with a diagnosis of heart failure with reduced or mildly reduced ejection fraction.

Inclusion Criteria:

* Patients aged 18 years and older
* Diagnosed with heart failure at the time of discharge
* Have an ejection fraction (based on imaging modalities such as echocardiography or cardiac MRI) recorded closest to the time of discharge, showing a left ventricular ejection fraction of less than 50%

Exclusion Criteria:

* Patients and their relatives do not have means of communication with healthcare staff (phone, computer, messaging, etc.)
* Patients do not reside in Vietnam after discharge

Data Collection:

* All patients meeting the criteria at the time of discharge during the study period will be continuously included. Information regarding demographic data, clinical presentation, biological markers, and in-hospital treatment characteristics will be collected using standardized data definitions from EuroHeart data standards for heart failure.
* Periodically after hospital discharge (e.g., 1 month, 3 months, 12 months post-discharge), patients will be contacted by investigators to gather information on their current status, medications, and any cardiovascular events, including rehospitalizations, death, and current medical treatment.
* Data entry will be performed using the REDCap project at the University of Medicine and Pharmacy, Ho Chi Minh City (https://redcap.umc.edu.vn/)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Diagnosed with heart failure at the time of discharge
* Have an ejection fraction (based on imaging modalities such as echocardiography or cardiac MRI) recorded closest to the time of discharge, showing a left ventricular ejection fraction of less than 50%

Exclusion Criteria:

* Patients and their relatives do not have means of communication with healthcare staff (phone, computer, messaging, etc.)
* Patients do not reside in Vietnam after discharge

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All eligible patients discharged with a diagnosis of heart failure with reduced or mildly reduced ejection fraction.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 12 months
  Death from any cause
Heart failure rehospitalization | 12 months
  Patient rehospitalization due to cardiovascular causes, excluding apparent non-cardiac causes.

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 12 months
  Acute myocardial infarction, stroke or death from any cause
Guideline-directed medical therapy detail | 12 months
  Information regarding guideline-directed medical therapy, including medications used and dose titration over time.

CONTACTS AND LOCATIONS:
Overall Officials: Cong Thanh Nguyen, MD, MSc, Study Chair — University Medical Center Ho Chi Minh City; Thanh Hai Nam Phan, MD, MSc, Study Chair — University Medical Center Ho Chi Minh City; Quang Binh Truong, Professor, Study Director — University of Medicine and Pharmacy at Ho Chi Minh City; Hoang Vu Vu, PhD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City; Dang Duy Quang Pham, MD, MSc, Study Chair — University Medical Center Ho Chi Minh City
Locations (1):
- University Medical Center Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Result] Aktaa S, Batra G, Cleland JGF, Coats A, Lund LH, McDonagh T, Rosano G, Seferovic P, Vasko P, Wallentin L, Maggioni AP, Casadei B, Gale CP; Heart Failure Association of the European Society of Cardiology. Data standards for heart failure: the European Unified Registries for Heart Care Evaluation and Randomized Trials (EuroHeart). Eur Heart J. 2022 Jun 14;43(23):2185-2195. doi: 10.1093/eurheartj/ehac151. PMID 35443059